CLINICAL TRIAL: NCT04198311
Title: The Impact of CBT for Insomnia on Substance Use Treatment Outcomes
Brief Title: Sleep Treatment for Addiction Recovery
Acronym: STAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Mary E Miller, Professor, Psychiatry, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016896
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-03

CONDITIONS: Insomnia; Alcohol Use Disorder; Substance Use Disorders
Keywords: sleep; alcohol; drinking; insomnia; outpatient; inpatient; drug use
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Alcoholism; Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will participate in sessions individual Cognitive Behavioral Therapy for Insomnia (CBT-I).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive-Behavioral Therapy for Insomnia (CBT-I) (Experimental): Individual Cognitive Behavioral Therapy for Insomnia (CBT-I) delivered once a week for five (5) weeks
  Interventions: Behavioral: CBT-I

INTERVENTIONS:
Behavioral: CBT-I — CBT-I will be delivered individually, in five weekly sessions. Intervention components include sleep hygiene, sleep restriction, stimulus control, relaxation, cognitive therapy.
  Other Names: Cognitive-Behavioral Therapy for Insomnia

SUMMARY:
Project STAR aims to examine the feasibility, acceptability, and initial efficacy of a CBT-I supplement to outpatient alcohol and substance use treatment.

DETAILED DESCRIPTION:
Among those who receive treatment for alcohol use disorder (AUD), one in three relapses to problematic drinking within one year of treatment. Thus, additional treatment strategies are needed. Notably, up to 74% of individuals seeking treatment for AUD report co-occurring symptoms of insomnia, while 85% of those seeking SUD treatment report insomnia symptoms. Given the negative impact of insomnia on attention and emotion regulation, insomnia symptoms may decrease patients' abilities to attend to treatment for substance use and manage negative emotions that lead to craving and relapse. This project aims to examine the feasibility, acceptability, and initial efficacy of a CBT-I supplement to substance use treatment. Forty adults who meet diagnostic criteria for AUD or SUD and Insomnia Disorder will receive Cognitive Behavioral Therapy for Insomnia (CBT-I). In order to generate hypotheses regarding the efficacy of CBT-I for individuals who are and are not engaged in substance use treatment, we aim to recruit 20 participants who are engaged in substance use treatment through the community at baseline and 20 participants who are not. Outcomes will be assessed at the end of the active intervention period (6 weeks) and at 6 weeks post-intervention

ELIGIBILITY:
Inclusion Criteria:

* Participation in alcohol or substance use treatment in the Columbia, MO area
* DSM-5 criteria for moderate to severe Alcohol Use Disorder of Substance Use Disorder
* DSM-5 episodic criterion (duration at least 1 month) for Insomnia Disorder

Exclusion Criteria:

* unable to provide informed consent
* cognitive impairment
* continuous sobriety for 2+ months at baseline
* untreated sleep disorder requiring more than behavioral treatment for insomnia
* severe psychiatric disorder that requires immediate clinical attention
* initiation of a sleep medication in the past six (6) weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Assessed at Post-Treatment (week 6)
  The number of participants who complete baseline.
Retention | Assessed at Post-Treatment (week 6)
  The number of participants who complete all treatment sessions
Treatment Satisfaction | Assessed at Post-Treatment (week 6)
  The satisfaction rating participants give the treatment.Assessed using the Client Satisfaction Questionnaire; The Client Satisfaction Questionnaire is an 8-item measure of satisfaction with treatment that has been validated in substance use treatment settings. Items are scores from 1 to 4, with higher scores indicating greater satisfaction with treatment.

SECONDARY OUTCOMES:
Abstinence | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  The percentage of days during the past 6 weeks that the participant is abstinent from their drug of choice (alcohol or other substance). Assessed using the Timeline Followback (TLFB); TLFB allows participants to trace their alcohol and drug use back 42 days.
Heavy-Drinking Days | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  The percentage of days during the past 6 weeks that the participant engages in heavy drinking (>4/5 drinks/day for women/men). Assessed using the Timeline Followback (TLFB) for alcohol; TLFB allows participants to trace their alcohol use back 42 days.
Substance Use Days | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  The percentage of days during the past 6 weeks that the participant engages in drug/substance use. Assessed using the Timeline Followback (TLFB) ; TLFB allows participants to trace their drug/substance use back 42 days.
Alcohol Problems | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  Assessed using the Short Inventory of Problems (SIP); SIP measures adverse consequences of substance use.
Alcohol or Other Drugs as Sleep Aids | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  Assessed using the daily sleep diary; Sleep Diaries are quotidian questionnaires that measure self-reported sleep quality, sleep time, and daily habits concerning substance use. Diaries will be used to determine if participants used alcohol or other substances specifically to go to sleep
Insomnia severity | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  Assessed using the Insomnia Severity Index (ISI); ISI will be used as a 7-item measure of insomnia severity in the past two weeks. Items assess difficulty falling or staying asleep, satisfaction with current sleep pattern, interference with daily functioning, the extent to which others notice their sleep problems, and worry/distress related to sleep problems. Response options range from 0 (not at all worried) to 4 (very much worried), with possible total scores ranging from 0 to 28. Participants scoring 10 or higher will be classified as screening positive for insomnia (Morin et al., 2011).114 Notably, self-report is the recommended method of assessment for symptoms of insomnia in adults (Schutte-Rodin et al., 2008).
Total Wake Time | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  The amount of time the participant is awake after they try to go to sleep. Measured using Daily Diaries and actigraphy.
Sleep quality | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  Assessed using the daily sleep diary; Sleep Diaries are quotidian questionnaires that measure self-reported sleep quality, sleep time, and daily habits concerning substance use. Diaries will be used to determine if participants used alcohol or other substances specifically to go to sleep.
Dysfunctional beliefs | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  Assessed using the Dysfunctional Beliefs and Attitudes about Sleep questionnaire (DBAS;Morin, 1994). The DBAS is designed to measure sleep and insomnia-related cognitions.

OTHER OUTCOMES:
Treatment-related Learning | Change from baseline to post-treatment (week 6)
  Assessed using the Project STAR alcohol quiz
Executive Functioning - Delayed Discounting | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  Assessed delayed discounting using the Monetary Choice Questionnaire (Kirby, Petry, & Bickel, 1999). Participants are instructed to choose between hypothetically receiving one amount of money today or a larger amount of money in the future.
Executive Functioning - Working Memory | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  Assessed using the Adaptive N-Back task (Jaeggi et al., 2010).Participants are instructed to indicate if the image they see is the same shape that was presented earlier.
Executive Functioning - Attention | Change from baseline to post-treatment (week 6) to follow-up (week 12)
  Assessed using the Psycho-motor Vigilance Task (Thomann et al., 2014). Participants are instructed to react to a visual stimulus by quickly pressing a key.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

REFERENCES:
- [Derived] Miller MB, Freeman LK, Helle AC, Hall NA, DiBello AM, McCrae CS. Comparative feasibility and preliminary efficacy of CBT for insomnia among adults seeking and not seeking addiction treatment. J Sleep Res. 2024 Apr;33(2):e13969. doi: 10.1111/jsr.13969. Epub 2023 Jul 9. PMID 37423902